CLINICAL TRIAL: NCT07000201
Title: the Sedative Efficacy of Preoperative Pregablin Versus Gabapentin in Elderly Undergoing Abdominopelvic Surgery : a Randomized Controlled Clinical Trial
Brief Title: Preoperative Pregabalin vs Gabapentin in Elderly Undergoing Surgry,Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marianne Magdy Youssef, Lecturer of anaesthesia ,icu & pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N-70-2025
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Anxiety Disorder (Panic Disorder or GAD)
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group I patients will receive two capsules of pregabalin (Lyrica) 75 mg (total = 150 mg), (Active Comparator)
  Interventions: Drug: One hour prior to admission to the operating room, patients will receive the study medication (as premedication) by mouth with a sip of water;
- group II patients will receive two capsules of gabapentin (Conventin) 300 mg (total = 600 mg), (Active Comparator)
  Interventions: Drug: One hour prior to admission to the operating room, patients will receive the study medication (as premedication) by mouth with a sip of water;
- group III patients will receive a matching placebo in the form of two capsules of powdered multivita (Placebo Comparator)
  Interventions: Drug: One hour prior to admission to the operating room, patients will receive the study medication (as premedication) by mouth with a sip of water;

INTERVENTIONS:
Drug: One hour prior to admission to the operating room, patients will receive the study medication (as premedication) by mouth with a sip of water; — group I patients will receive two capsules of pregabalin (Lyrica) 75 mg (total = 150 mg), group II patients will receive two capsules of gabapentin (Conventin) 300 mg (total = 600 mg), and group III patients will receive a matching placebo in the form of two capsules of powdered multivitamin by mouth.

SUMMARY:
Several studies have evaluated the efficacy of pregabalin in reducing preoperative anxiety, with inconsistent results. Similarly, inconclusive results have been reported regarding gabapentin and its effects in reducing preoperative anxiety. A previous study reported that a single dose of gabapentin or pregabalin administered 60 minutes before surgery in adults under general anesthesia was effective in reducing acute preoperative anxiety and elevated levels of sedation before and after surgery, with pregabalin having better anxiolytic and sedative effects than gabapentin. However, no previous studies have compared the efficacy of preoperative pregabalin or gabapentin as premedication to reduce intraoperative anxiety and induce sedation in geriatric patients undergoing major surgery with regional anesthesia

ELIGIBILITY:
Inclusion Criteria:This study will include :

1. geriatric patients, aged 65 years or older,
2. Both sex,
3. scheduled for elective abdominopelvic surgery with regional anesthesia
4. American Society of Anesthesiologists (ASA) physical status I or II.

Exclusion Criteria:We will exclude patients with any of the following:

1. history of allergy to gabapentin or pregabalin;
2. current use of gabapentin or pregabalin for other indications
3. history of chronic pain or chronic daily use of analgesics; a
4. history of epilepsy, other neurological disorders, cognitive impairment, or severe psychiatric disorders;
5. severe cardiovascular or respiratory diseases;
6. impaired renal function; and a history of drug or alcohol abuse.
7. patients with anticipated prolonged duration of surgery for more than two hours

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative sedation levels are assessed using the Ramsay Sedation Scale . | 1 hour after giving the drug
  The Ramsay Sedation Score is a scale used to assess the level of sedation in patients. It ranges from 1 to 6, with higher scores indicating a deeper level of sedation score 1: Patient is anxious, agitated, or restless. Score 2: Patient is cooperative, oriented, and tranquil. Score 3: Patient responds to commands only. Score 4: Patient responds briskly to a light glabellar tap or loud auditory stimulus.
  Score 5: Patient responds sluggishly to a light glabellar tap or loud auditory stimulus.
  Score 6: Patient does not respond to pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralaini medical school, Cairo, Giza Governorate, Egypt